CLINICAL TRIAL: NCT00994565
Title: The Effectiveness of Physical Activity Monitoring and Distance Counselling in an Occupational Health Setting - a Randomised Controlled Trial (CoAct)
Brief Title: The Effectiveness of Physical Activity Monitoring and Distance Counseling in an Occupational Health Setting
Acronym: CoAct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University of Technology (Other)
Collaborators: The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government); Pohjola Insurance Ltd (Unknown)
Responsible Party: Simo P. Taimela / MD, PhD., Department of Public Health, Helsinki University
Organization: HelsinkiUT (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CoAct1RCT
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Physical Inactivity
Keywords: Physical activity; health behaviour; lifestyle; productivity; outcomes
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Distance Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention)
- Activity monitoring and distance counseling (Active Comparator)
  Interventions: Behavioral: Activity monitoring and distance counseling

INTERVENTIONS:
Behavioral: Activity monitoring and distance counseling — The physical activity monitoring and distance counseling concept combines the use of a personal activity monitor with web-based tailored physical activity advice. Users can interactively plan and evaluate their own activity advice based on their actual PA scores and their PA preferences and goals.
  Arms: Activity monitoring and distance counseling

SUMMARY:
The CoAct study is investigating a novel lifestyle intervention, aimed at the working population, with daily activity monitoring and distance counseling via telephone and secure web messages. The main purpose of this study is to evaluate the effectiveness of lifestyle counseling on the level of physical activity in an occupational health setting. The purposes include also analyzing the potential effects of changes in physical activity on productivity at work and sickness absence, and health care costs.

DETAILED DESCRIPTION:
CoAct is a randomized controlled trial with two arms: a control group and intervention group with daily activity monitoring and distance counseling. The intervention focuses on lifestyle modification and takes 12 months. The study population consists of those volunteering from 1100 eligible employees from a Finnish insurance company. The primary outcomes are change in physical activity measured in MET hours per week, work productivity and sickness absence, and health care utilization. Secondary outcomes include various physiological measures. Cost-effectiveness analysis will also be performed. The outcomes will be measured by questionnaires at baseline, after 6, 12, and 24 months, and sickness absence will be obtained from the employer's registers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Paid employment of at least 8 hours a week
* Not scheduled to retire in the next two years or have applied for disability pension
* Have completed a health risk appraisal and physical testing

Exclusion Criteria:

* Pregnancy
* Diagnosis or treatment of cancer
* Any disorder that makes physical activity impossible

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 544 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Physical Activity | One year

SECONDARY OUTCOMES:
Health related productivity loss | One year
Healthcare utilization | One Year

CONTACTS AND LOCATIONS:
Locations (1):
- BIT Research Center, Espoo, Finland

REFERENCES:
- [Derived] Reijonsaari K, Vehtari A, Kahilakoski OP, van Mechelen W, Aro T, Taimela S. The effectiveness of physical activity monitoring and distance counseling in an occupational setting - results from a randomized controlled trial (CoAct). BMC Public Health. 2012 May 11;12:344. doi: 10.1186/1471-2458-12-344. PMID 22578104
- [Derived] Reijonsaari K, Vehtari A, van Mechelen W, Aro T, Taimela S. The effectiveness of physical activity monitoring and distance counselling in an occupational health setting--a research protocol for a randomised controlled trial (CoAct). BMC Public Health. 2009 Dec 31;9:494. doi: 10.1186/1471-2458-9-494. PMID 20043831